CLINICAL TRIAL: NCT07343505
Title: A Prospective Study Investigating the Effects of an Environmental Enrichment-Based Intervention on Brain Development in Preterm Infants
Brief Title: Environmental Enrichment Intervention and Brain Development in Preterm Infants
Acronym: PRE-ENV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Tuğçe Altıok, PhD Candidate, Eskisehir Osmangazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESOGU-TA-PretermEE-001; TDK-2025-3575 (Other Grant/Funding Number: Scientific Research Projects (BAP), Eskisehir Osmangazi University)
Record Dates: First submitted 2025-11-21; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth
Keywords: Preterm infants; Environmental enrichment; Home-based intervention; Early intervention; Brain development; Cognitive development; Motor development; Neurodevelopment
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Participants will be prospectively assigned to one of two parallel groups using stratified assignment based on gestational age. One group will receive standard care alone, while the other group will receive a structured environmental enrichment-based HEP home intervention in addition to standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Infants in this group will receive conventional developmental therapy and routine medical follow-up as provided within standard clinical practice. This approach represents an active comparator and does not include the structured environmental enrichment or the Homeostasis-Enrichment-Plasticity (HEP)-based intervention used in the experimental group. Participants in this group will undergo the same study-related assessments as the intervention group at baseline and after 12 weeks.
  Interventions: Other: Standard Developmental Care
- HEP Home-Practice Group: (Experimental): A structured environmental enrichment-based developmental intervention delivered over a 12-week period. The program is based on the Homeostasis-Enrichment-Plasticity (HEP) framework and includes age-appropriate sensory-motor activities, environmental novelty, problem-solving opportunities, and active caregiver-infant interaction. The intervention is delivered through weekly therapist-guided sessions, with caregivers encouraged to continue the practices at home as part of daily care.
  Interventions: Behavioral: Environmental Enrichment-Based Intervention

INTERVENTIONS:
Other: Standard Developmental Care — Standard developmental care and routine medical follow-up provided within usual clinical practice. This care reflects established developmental support approaches typically offered to preterm infants and does not include structured environmental enrichment or the Homeostasis-Enrichment-Plasticity (HEP)-based intervention applied in the experimental group.
  Arms: Control Group
Behavioral: Environmental Enrichment-Based Intervention — Environmental enrichment-based program applied for 12 weeks, including sensory-motor stimulation, environmental novelty, problem-solving tasks, and active exploration with caregivers.
  Arms: HEP Home-Practice Group:

SUMMARY:
This study aims to evaluate the effects of a structured environmental enrichment (EE)-based early developmental intervention on brain, motor, and cognitive outcomes in preterm infants. Infants born before 37 weeks of gestation are at increased risk for alterations in structural and functional brain development, which may be further influenced by the neonatal intensive care environment, including exposure to excessive light, noise, and frequent medical procedures.

The intervention is a prospectively implemented, home-based developmental program structured according to the HEP (Homeostasis-Enrichment-Plasticity) approach, providing enriched sensory-motor experiences, environmental novelty, problem-solving activities, and opportunities for active exploration. The program is delivered through guided parental involvement with support from trained therapists, according to a predefined protocol.

Developmental outcomes will be assessed at baseline and after the intervention period using standardized, non-invasive assessment tools. The intervention does not include any pharmacological treatment or medical device. This study evaluates whether participation in an EE-based early developmental intervention leads to improved neurodevelopmental outcomes in preterm infants.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of an environmental enrichment (EE)-based early developmental intervention on brain, motor, and cognitive development in preterm infants. Infants born before 37 weeks of gestation are at increased risk for alterations in brain structure and subsequent neurodevelopmental challenges. In addition to biological vulnerability, early sensory experiences and environmental factors may influence developmental trajectories during infancy.

This study will examine developmental outcomes together with brain morphometric measurements and urinary biochemical markers, including brain-derived neurotrophic factor (BDNF), nerve growth factor (NGF), Tau, and S100B.

Objectives:

1. To assess urinary biochemical markers, brain morphometry, and motor and cognitive development in preterm infants at corrected 1 month of age.
2. To examine relationships among urinary biochemical markers, brain morphometry, and developmental outcomes at baseline.
3. To compare changes in biochemical, neuroimaging, and developmental outcomes over a 12-week period between infants receiving standard care and those receiving an EE-based intervention.

Study Design:

A total of 28 preterm infants born before 37 weeks of gestation will be enrolled. The study will begin when infants reach corrected 1 month of age. Participants will be allocated into two parallel groups using stratified assignment based on relevant clinical characteristics.

Standard Care Group:

Infants in the standard care group will continue to receive routine medical follow-up and developmental monitoring as provided by their healthcare services. No additional intervention beyond usual care will be introduced as part of the study.

Environmental Enrichment (HEP) Intervention Group:

Infants in the intervention group will receive a structured environmental enrichment-based developmental program guided by a therapist through weekly in-person sessions. The intervention is based on the Homeostasis-Enrichment-Plasticity (HEP) approach and focuses on providing enriched sensory-motor experiences, environmental novelty, problem-solving opportunities, and active exploration appropriate to the infant's corrected age.

Weekly sessions are conducted by a trained therapist and are designed to support infant-environment interaction, promote motor and cognitive engagement, and coach caregivers in implementing developmentally appropriate practices. In addition to the therapist-guided sessions, caregivers are encouraged to integrate the HEP-based practices into their daily routines at home.

All intervention components are non-invasive, behavioral, and developmentally supportive in nature. No pharmacological treatments, invasive procedures, or medical devices are used as part of the intervention.

Procedures:

Urinary biochemical markers: Urine samples will be collected from all infants at baseline (corrected 1 month of age) and after the 12-week intervention period to measure levels of BDNF, NGF, Tau, and S100B. Samples will be stored at -80°C until analysis.

Brain imaging: Cranial ultrasonography obtained as part of routine clinical care will be used for morphometric analysis. No additional imaging procedures will be performed solely for research purposes.

Developmental assessment: Motor development will be assessed using the Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) Motor Scale and the Test of Infant Motor Performance (TIMP). Cognitive development will be evaluated using the Bayley-III Cognitive Scale.

Caregiver well-being: Caregivers will complete the Depression Anxiety Stress Scales-21 (DASS-21) to assess caregiver psychological status.

Follow-up and Analysis:

All outcome measures, including urinary biochemical markers, cranial ultrasonography, developmental assessments, and caregiver questionnaires, will be repeated after the 12-week intervention period. Statistical analyses will examine within- and between-group changes over time, as well as associations among biochemical markers, brain morphometry, and developmental outcomes.

ELIGIBILITY:
Inclusion Criteria

* Preterm infants born before 37 completed weeks of gestation.
* Corrected age between 4 and 7 weeks at the time of enrollment.
* Medically stable, as confirmed by the attending neonatologist
* Written informed consent obtained from parents or legal guardians.

Exclusion Criteria

* Major congenital anomalies or known genetic syndromes.
* Severe intraventricular hemorrhage (Grade III-IV) or other major neurological impairment.
* Unstable medical conditions that would interfere with safe participation in the study procedures.
* Caregivers unable to attend scheduled study sessions or comply with study-related procedures.

Ages: 4 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Motor Development Assessed by Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) | Baseline (corrected age of 1 month) and 12 weeks (end of intervention)
  Motor development will be assessed using the Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III), Motor Composite Score, which evaluates fine and gross motor development.
  The Motor Composite Score ranges from 40 to 160, with higher scores indicating better motor development.
Motor Performance Assessed by Test of Infant Motor Performance (TIMP) | Baseline (corrected age of 1 month) and 12 weeks (end of intervention)
  Motor performance will be assessed using the Test of Infant Motor Performance (TIMP), which evaluates postural and selective control of movement in young infants.
  The TIMP total score ranges from -49 to 142, with higher scores indicating better motor performance.

SECONDARY OUTCOMES:
Cognitive Development Assessed by Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) | Baseline (corrected age of 1 month) and 12 weeks (end of intervention)
  Cognitive development will be assessed using the Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III), Cognitive Composite Score, which evaluates cognitive abilities including attention, memory, and problem-solving.
  The Cognitive Composite Score ranges from 40 to 160, with higher scores indicating better cognitive development.
Brain Morphometric Measurements Assessed by Cranial Ultrasound Imaging | Baseline (corrected age of 1 month) and 12 weeks (end of intervention)
  Brain structural development will be evaluated using cranial ultrasound imaging with morphometric measurements, including ventricular size and selected linear brain dimensions.
  Changes in morphometric measurements over time will be used to assess brain structural development, with larger or more age-appropriate measurements indicating more advanced brain development.
Urinary Concentration of Brain-Derived Neurotrophic Factor (BDNF) | Baseline (corrected age of 1 month) and 12 weeks (end of intervention)
  Urine samples will be collected to measure the concentration of brain-derived neurotrophic factor (BDNF) using standardized immunoassay methods.
  BDNF levels will be reported as urinary concentration, and changes in concentration over time will be used to evaluate neurodevelopmental effects of the intervention.
  Higher BDNF levels indicate enhanced neurotrophic support.
Urinary Concentration of Nerve Growth Factor (NGF) | Baseline (corrected age of 1 month) and 12 weeks (end of intervention)
  Urine samples will be collected to measure the concentration of nerve growth factor (NGF) using standardized immunoassay methods.
  NGF levels will be reported as urinary concentration, and changes in concentration over time will be used to assess neurodevelopmental support.
  Higher NGF levels indicate enhanced neurodevelopmental processes.
Urinary Concentration of Tau Protein | Baseline (corrected age of 1 month) and 12 weeks (end of intervention)
  Urine samples will be collected to measure the concentration of Tau protein using standardized immunoassay methods.
  Tau levels will be reported as urinary concentration, and changes in concentration over time will be interpreted in relation to neuronal integrity.
  Alterations in Tau concentration may reflect changes in neuronal structure or injury.
Urinary Concentration of S100 Calcium-Binding Protein B (S100B) | Baseline (corrected age of 1 month) and 12 weeks (end of intervention)
  Urine samples will be collected to measure the concentration of S100 calcium-binding protein B (S100B) using standardized immunoassay methods.
  S100B levels will be reported as urinary concentration, and changes in concentration over time will be used to evaluate brain structural integrity.
  Elevated S100B levels are interpreted in relation to brain tissue stress or injury.
Depression, Anxiety, and Stress Scale-21 Items (DASS-21) Total and Subscale Scores in Caregivers | Baseline and 12 weeks (post-intervention)
  Caregiver psychological status will be assessed using the Depression, Anxiety, and Stress Scale-21 Items (DASS-21), a self-report questionnaire consisting of three subscales: depression, anxiety, and stress.
  Each subscale score ranges from 0 to 42, with higher scores indicating greater levels of depression, anxiety, or stress.
  Changes in total and subscale scores over time will be used to evaluate the psychological impact of the intervention on caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Altıok, PhD, Study Director — Eskisehir Osmangazi University, Institute of Health Sciences; Ferruh Yücel, Professor, PhD, Principal Investigator — Eskisehir Osmangazi University; Aymen Balıkçı, PT, PhD, Study Director — Aymen Balıkçı Physical Therapy Clinic; Teresa A. May-Benson, PhD, Study Director — Teresa A. May-Benson Therapy Clinic
Locations (1):
- Tuğçe Altıok Physical Therapy Center, Nilufer, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.